CLINICAL TRIAL: NCT04706013
Title: Study of Pyridoxal 5'-Phosphate for the Treatment of Patients With PNPO Deficiency
Brief Title: Oral Pyridoxal 5'-Phosphate for the Treatment of Patients With PNPO Deficiency
Acronym: MEND-PNPO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Medicure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEND-PNPO 16002
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Pyridox(am)Ine 5'-Phosphate Oxidase Deficiency
MeSH Terms: interventions — Pyridoxal Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm Active (Experimental): Pyridoxal 5'-Phosphate
  Interventions: Drug: Pyridoxal Phosphate

INTERVENTIONS:
Drug: Pyridoxal Phosphate — Oral tablets 50 mg

SUMMARY:
The proposed clinical study is intended to evaluate oral P5P for the treatment of patients confirmed to have Pyridox(am)ine 5'-Phosphate Oxidase (PNPO) deficiency via genetic analysis. There is an unmet clinical need for pharmaceutical grade P5P, as to date none has been made commercially available. Patients will receive pharmaceutical grade P5P according to their normal oral P5P dosing regimen, as previously established by their physicians.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed PNPO deficiency via genetic analysis, whose seizures are typically controlled on P5P (oral) therapy.

   a. Typically controlled is defined as receiving multiple doses of P5P daily to control seizures. Receiving P5P for a minimum of 30 days.
2. Male and/or female patients.
3. Aged ≥2 years

(3) Patients with previous failed treatment on pyridoxine are eligible for the study (patient should be off pyridoxine for at least 24 hours).

(4) Written informed consent (by parent or guardian if under the age of 18).

Exclusion Criteria:

1. The patient has any condition or abnormality which may, in the opinion of the Investigator, compromise the safety of the patient, or influence their ability to comply with study procedures.
2. Known or suspected allergy to the trial drug or the relevant drugs given in the trial.
3. Involvement in a clinical research study within 4 weeks prior to screening and/or prior enrollment in the study. Participation in observational registry studies is permitted.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival time (time to death), including incidence of death at 12 months | 12 months
  The study group will be compared to a historical control group (without active treatment) for overall survival by using the method of survival analysis

SECONDARY OUTCOMES:
Frequency of seizures (including but not limited to status epilepticus) | up to 12 months
  The frequency of seize will be compared between different treatment periods of the current single arm: Pharmaceutical grade oral P5P treatment period vs period prior to any P5P treatment (if data available)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke Children's Hospital, Durham, North Carolina
  - Akron's Children's Hospital, Akron, Ohio
- Queensland Children's Hospital, South Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided